CLINICAL TRIAL: NCT00000755
Title: A Phase I/II Trial of Vaccine Therapy of HIV-1 Infected Individuals With 50-500 CD4 Cells/mm3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: ACTG 209; 11186 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; HIV Envelope Protein gp120; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Biological: rgp120/HIV-1MN
Drug: Zidovudine

SUMMARY:
To examine the response of HIV-1 infected patients to vaccination with gp120/HIV-1MN antigen. To determine the effect of antiretroviral therapy on vaccine responsiveness.

Fifty percent of HIV-1 infected individuals remain symptom free for 8-12 years. It has been hypothesized that HIV-specific immune responses are responsible for the period of relative quiescence of viral replication. Recent studies suggest that these immune functions can be augmented by vaccination with HIV-derived antigens.

DETAILED DESCRIPTION:
Fifty percent of HIV-1 infected individuals remain symptom free for 8-12 years. It has been hypothesized that HIV-specific immune responses are responsible for the period of relative quiescence of viral replication. Recent studies suggest that these immune functions can be augmented by vaccination with HIV-derived antigens.

Patients are randomized to receive rgp120/HIV-1MN vaccine or alum adjuvant placebo by intramuscular injection at weeks 0, 4, 8, 12, 16, and 20, with or without daily oral zidovudine (AZT) or their current stable dose of antiretroviral therapy. After completing the primary vaccination series, patients are permitted to continue into an extension phase, in which they receive a booster vaccination at weeks 28, 36, and 44. Patients will be stratified by CD4 count: 350-500, 200-349, and 50-199 cells/mm3. A fourth group with counts of 350-500 cells/mm3 will serve as a pilot group and receive vaccine only.

ELIGIBILITY:
Inclusion Criteria

Required immediately prior to study entry:

* A minimum of 2 and a maximum of 12 months of AZT therapy at 500-600 mg/day (does not apply to the pilot group patients receiving vaccine only and to patients with CD4 counts of 50-199 cells/mm3).

Concurrent Medication:

Allowed:

* PCP prophylaxis.
* Rifabutin and clarithromycin (in patients with CD4 counts of 50-199 cells/mm3 only).
* Short-term nonsteroidal anti-inflammatory therapy for acute conditions.
* Short intermittent cycles of acyclovir.

Patients must have:

* HIV infection, with CD4 count of 50-500 cells/mm3.
* No active opportunistic infection (patients with CD4 counts of 50-199 cells/mm3 may have a history of an opportunistic infection).
* Consent of parent, guardian, or person with power of attorney, if less than 18 years of age.
* B-cell lines established in order to be vaccinated.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known or suspected allergies to any vaccine components.

Concurrent Medication:

Excluded:

* Agents with immunosuppressive activity.
* Antiretroviral therapies other than AZT (except in patients with CD4 counts of 50-199 cells/mm3).
* Interferon.
* Parenteral therapies (including SC allergy medications and chemotherapy for Kaposi's sarcoma).
* Steroids.
* Hematopoietins.

Prior Medication:

Excluded within 12 weeks prior to study entry:

* Agents with immunosuppressive activity.
* Antiretroviral therapies other than AZT (except in patients with CD4 counts of 50-349 cells/mm3).
* Interferon.
* Parenteral therapies (including SC allergy medications and chemotherapy for Kaposi's sarcoma).
* Steroids.
* Hematopoietins.

Active drug abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168
Dates: Study Completion 1993-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Schooley RT, Study Chair; Walker B, Study Chair
Locations (10):
- United States (10):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - NY Univ. HIV/AIDS CRS, New York, New York
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Kuritzkes DR, Spino C, Valentine F, Schooley RT. Association of plasma HIV-1 RNA, CD4 count, and immune response in patients with 50-500 CD4 cells/ul. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:204 (abstract no 757)
- [Background] Schooley RT, Spino C, Chiu S, DeGruttola V, Kuritzkes DR. Poor immunogenicity of HIV-1 envelope vaccines with alum or MF59 aduvant in HIV-infected individuals: results of two randomized trials. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:204 (abstract no 756)
- [Background] Schooley RT, Spino C, Kuritzkes D, Walker BD, Valentine FA, Hirsch MS, Cooney E, Friedland G, Kundu S, Merigan TC Jr, McElrath MJ, Collier A, Plaeger S, Mitsuyasu R, Kahn J, Haslett P, Uherova P, deGruttola V, Chiu S, Zhang B, Jones G, Bell D, Ketter N, Twadell T, Chernoff D, Rosandich M. Two double-blinded, randomized, comparative trials of 4 human immunodeficiency virus type 1 (HIV-1) envelope vaccines in HIV-1-infected individuals across a spectrum of disease severity: AIDS Clinical Trials Groups 209 and 214. J Infect Dis. 2000 Nov;182(5):1357-64. doi: 10.1086/315860. Epub 2000 Oct 9. PMID 11023459